CLINICAL TRIAL: NCT05121753
Title: Infant Formula Feeding and the Etiology of Necrotizing Enterocolitis in Newborns Survey
Brief Title: Infant Formula Feeding and Necrotizing Enterocolitis in Newborns
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuroganics LLC (Industry)
Collaborators: Ramos Law Injury Firm (Unknown)
Responsible Party: Sponsor
Other Study IDs: NEC_1121
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Necrotizing Enterocolitis; Necrotizing Enterocolitis of Newborn; Sepsis Newborn; Cows Milk Allergy
MeSH Terms: conditions — Enterocolitis, Necrotizing; Neonatal Sepsis; Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

INTERVENTIONS:
Dietary Supplement: Survey investigating Infant formula feeding in newborns — A database will be created that allows individuals to register and enter information about the premature infant's feeding history and symptoms/ medical history.

SUMMARY:
Necrotizing enterocolitis (NEC) is the most common life-threatening gastrointestinal emergency of prematurity, associated with a significant morbidity and mortality. Early diagnosis and early treatment interventions may reduce the risk of mortality and morbidity.

The Primary goal of this observational study is to gather survey data to establish a national database of NEC in newborns in order to better understand the risk factors underlying NEC. Survey data will be used along with a medical history to identify the mechanism(s) underlying the increased prevalence of NEC in non-breast fed, formula fed premature infants.

DETAILED DESCRIPTION:
NEC affects between 2 to 7% of premature infants. It is is an acquired disease, caused, in part by inflammation of the intestinal lining. NEC is the most common life-threatening gastrointestinal emergency of prematurity and it is associated with significant morbidity and mortality.

Studies have linked the consumption of non-breast milk, commercial infant formula (made from cow's milk) or formula-derived nutrition with increased risk of NEC compared to consumption of human breast milk.

The mechanism of the NEC lesions appears to involve factors including allergic reaction to the infant formulas containing cow's milk, immaturity of the intestinal barrier and the immune system, microvascular imbalance, disturbed gut flora and systemic inflammation that is hypothesized to be exacerbated by infant formula consumption.

The primary goal of this National observational study is to gather survey data in order to establish a database of NEC in newborns to gain a better understanding of the risk factors underlying NEC. Survey data will be used along with a medical history to identify the mechanism(s) underlying the increased prevalence of NEC in non-breast fed, formula fed premature infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants born after 2018
* Newborns that have been diagnosed with NEC and have consumed infant formula.
* Infants whose death resulted from NEC or complications thereof

Exclusion Criteria:

* Infants who were born prior to 2019
* Newborns who have been fed exclusively on breast milk.
* Subjects lacking medical records or who cannot provide a medical history.

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn infants fed formula and experienced symptoms of NEC.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Infant formulas and increased risk for NEC survey | 2 years
  A survey is given to allow parents/ guardians or health care workers to describe the events leading up to the development of NEC in their newborn.

CONTACTS AND LOCATIONS:
Overall Officials: Don Cooper, Ph.D., Principal Investigator — Neuroganics LLC
Locations (1):
- 10190 Bannock St #102, Northglenn, Colorado, United States